CLINICAL TRIAL: NCT03993860
Title: Introduction of Fish Early in the Complementary Feeding Period to Improve Infant Growth in Samfya District, Luapula Province, Zambia
Brief Title: Introduction of Fish Early in the Complementary Feeding Period to Improve Infant Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mukuba University (Other)
Collaborators: University of Stellenbosch (Other); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Given Chipili, Principal Investigator, Mukuba University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STC/2019/03
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Infant Growth
Keywords: Infants; Growth; Stunting; Fish; Intervention
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Intervention Model Description: An independent statistician not be part of the study prepared the randomisation schedule. All eligible infants were randomly assigned to either the intervention (Chisense fish powder) or the control (placebo in the form of sorghum powder) group at 6 months. A 1:1 ratio using a computerised random number generator and block randomisation in Microsoft Excel was used to randomise the infants to two groups of equal size. The schedule was stratified by the gender of infants (boy or girl) to enable gender balance in both groups. Allocation of concealment was done using a central randomisation service through a computer algorithm to protect the randomisation schedule. If there two infants from the same household or in case of twins, they were treated as a single baby during randomisation to avoid contamination. However, each child had his or her own code and will be assessed as an individual throughout the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: During grinding of sorghum powder, roasted small fish (3g/100g of sorghum) was added to the sorghum to provide a similar fish aroma as the fish product. The fish powder (12g)/ sorghum powder (12g) was then pre-packed in small plastic sachets. The participant and the field workers (research assistants and health workers) are blinded while the principal investigator (PI) is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Infants will be given fish powder called Chisense (Potamothrissa acutirostris) for a period of 6 months from the time they are 6 months up to the time they are 12 months.
  Interventions: Dietary Supplement: Fish Powder
- Control arm (Placebo Comparator): Infants will be given fish powder called sorghum powder for a period of 6 months from the time they are 6 months up to the time they are 12 months.
  Interventions: Dietary Supplement: Sorghum powder

INTERVENTIONS:
Dietary Supplement: Fish Powder — Dry small fish (Chisense) is roasted and ground into a powder and packed in a sachet (12g) and given to the child at 6 months up to the time the child is 12 moths old. Each month the childs anthropometric measurement are taken to monitor growth.
  Arms: Intervention arm
Dietary Supplement: Sorghum powder — Dry sorghum is roasted and ground into a powder and packed in a sachet (12g) and given to the child at 6 months up to the time the child is 12 moths old. Each month the childs anthropometric measurement are taken to monitor growth.
  Arms: Control arm

SUMMARY:
The aim of the study is to provide proof that giving fish during early complementary feeding improves infant linear growth outcomes.

DETAILED DESCRIPTION:
Stunting is an irreversible consequence of inadequate growth during the early life of a child in the absence of appropriate interventions before the age of 2 years. Stunting affect 151 million (22.2%) of children worldwide. World Health Organisation (WHO) global nutrition target for 2025 is to reduce the number of stunted children under-five years by 40%.3,4 The first 1000 days (conception to 2years) is crucial for later development. It is also the period when stunting prevalence is at its highest. In Zambia, the stunting prevalence is 40%8 , 43% in Luapula province with Samfya district statistics as high as 49%.

Good complementary feeding of children contributes to the positive characteristics of growth trends observed in developed countries. It is a period of introducing solids and age of accelerated growth. Improved linear growth in food insecure homes is achievable by using locally available foods that are sustainable and usually acceptable. The role of fish's contribution to child's optimal growth and development in the first 1 000 days in Zambia has been reviewed. A food consumption survey also shows that fish is one of the highly consumed protein foods in low-income households in Zambia.To the investigators knowledge, fish has not been assessed as an early complementary food for infants aged 6 months in Zambia. This study will investigate the effect of providing dry fish powder to 6 months old infants (over a 6 months period) on their linear growth Research Question Can the introduction of fish during early complementary feeding improve infant linear growth in Samfya district, Zambia? Study Aim The aim of this study is to determine if the introduction of fish during early complementary feeding improves infant's linear growth outcomes.

Objectives Primary Objective The primary objective of the study is to evaluate the effect of introducing fish during early complementary feeding on growth outcomes of infants in Samfya district, Zambia.

Secondary Objectives

* To determine the prevalence of stunting in 6-months old children in the study area.
* To determine the prevalence of stunting in 6-months old children in the study area.
* To determine basic and underlying (socio-demographic, infants/maternal history) factors associated with stunting, wasting and underweight in the study area
* To determine the prevalence of fish allergy in the study area
* To assess the acceptability of fish powder as an early complementary food.

Methodology

Samfya district is a rural area in North-East Zambia in Luapula Province and has 210, 251 inhabitants, of which 42, 050 (20%) are under-five children. The study will be conducted at Shikamushile Rural Health Centre (RHC) in Samfya district. Shikamushi RHC is one of the 10 RHCs without any nutrition programme. It serves a population of 11, 800; 2400 (20%) of these children attend the under-five clinic at the centre. This centre has more cases of malnourished children referred to the hospital for treatment than any other RHC.

The study will be a single blinded randomised controlled trial. The trial will have two arms with the intervention group receiving fish powder (Chisense) while the control will be given a placebo in the form of sorghum powder. Infants aged 6 months will be followed up for a period of 6 months until they are 12 months old. The total sample size estimate is 238 infants, 119 infants per group with the possible attrition rate of 20%, and power of 80% to detect a 0.45 growth difference in length-for-age Z score between the intervention and control group.

The investigator intends to use a questionnaire to collect socio-demographic data and take anthropometric measurements (from both mothers and infants) at baseline to determine basic and underlying factors associated with stunting, wasting and underweight in the study area. The data set will include, mother's age, nutrition status, number of births, source of drinking water, family size, source of income, breastfeeding and complementary food. Anthropometric measurements will be used to determine the prevalence of stunting, wasting and underweight in the study area. In addition, a 24-hour dietary recall questionnaire will be administered to determine the type of food given to children. Furthermore, a skin prick test will be conducted at baseline on infants aged 6 months to determine the prevalence of fish allergy in the study area.

Infants will then be followed up for 6 months during which, infants in the intervention group will receive 12g (7.6g protein) fish powder while the control will receive 7g (0.9g protein) sorghum powder per day. The follow-up will include, weekly and monthly follow-up Weekly home visits: During weekly home visits, the research assistants will distribute pre-packed fish/sorghum powder to last a week to the intervention and control group respectively. Research assistants will keep record of any morbidities experienced by the infants. Adherence to the intervention will be assessed by reports from mothers of infants and empty fish powder storage bowls.

Monthly RHC visits: Each month the mothers in both the intervention and control group will have their infant's anthropometric (weight, length, head circumference and mid-upper aim circumference) measurements taken during visits at the RHC. A 24-hour dietary recall will be administered every two months to determine dietary intake of infants. After the intervention, mothers of infants will be given a questionnaire to assess acceptability of fish as an early complementary food. The questionnaire will have questions on the flavour, colour, and consumption.

Statistical Analysis: Descriptive statistics will be used to describe the incidence of allergy among the study infants. The relationships between continuous response variables and nominal input variables, for example different diets, will be analysed using appropriate ANOVA or pooled or Welch t-tests if the two groups are involved. Appropriate repeated measures ANOVA will be used when responses are measured at specific time intervals. When only two times are compared, this will be done with paired t-tests. The relation between nominal variables will be investigated with contingency tables and appropriate chi-square tests, such as the likelihood ratio chi-square test. A p-value of p < 0.05 will represent statistical significance and 95% confidence intervals will be used to describe the estimation of unknown parameters.

The study protocol has approval from the Health Research Ethics Committee (HREC) and Tropical Disease Research Centre (TDRC), Ndola Zambia. . Permission to conduct the study at Sikamushile rural health center was sought from Samfya District Medical Office (SDMO). The following was ensured, informed consents, freedom of participation/withdrawal, and anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 6 months attending under-five clinic at the sampled RHC. Infants should ideally be 6 months of age however, the study will provide leeway of 2 weeks, and therefore infants falling within the age range 5.5 - 6.5 months may be included. If a 5.5-month-old infant has however not been started with complementary food, the mother will be advised to only start at the age of 6 months with the product.
* Infants whose mothers give written consent
* Infants whose mothers have no plans of moving away during the study period

Exclusion Criteria:

* Infants with, chronic or congenital diseases/disorders that may affect the growth of the children. These may include Down syndrome, cerebral palsy, spina bifida and any other related condition.
* Premature infants
* infected infants

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Linear growth | At baseline (6 months), 7,8,9,10,11 and 12 months.
  Mean change from baseline in length-for-age Z-scores at 7, 8, 9,10,11 and 12 months old.:WHO 2006 Growth Standards

SECONDARY OUTCOMES:
The percentage (%) of infants who will be stunted. | At baseline (6 months) 7, 8, 9,10,11 and 12 months
  Mean length-for-age Z-scores at baseline (6 months), 7, 8, 9,10,11 and 12 months : WHO 2006 Growth Standards
The percentages (%) of infants who will be underweight and wasted in the study. | At baseline (6 months) 7, 8, 9,10,11 and 12 months
  Mean Weight-for-length/Weight-for_age at baseline (6 months) for-age WHO 2006 growth Standards.
The percentage (%) of infants who will be allergic to fish . | 6 months
  A skin prick test using fish (chisense) extract. Histamine dihydrochloride 10 mg/ml as a positive and water as a negative control. A skin reaction of more than 3mm will be considered positive.
Acceptability of fish powder as an early complementary food: | At end-line of the study (when infants are 12 months old)
  Mothers of infants in the intervention group will be interviewed on the acceptability of fish as an early complementary food using a questionnaire. Taste, smell, colour, flavour, amount consumed by the infant (grams per day). Fours (4) scores out of five (5) will be considered acceptable.
Factors associated with stunting, wasting and underweight in the study area. | After collecting baseline information (When infants are 6 months old)
  The socio-demographic data ( for example; age of the mother, level of education, occupation, family size, source of income and marital status) will be compared with the results of the infant's anthropometric measurements. Linear regression mixed effect regression modal will be used to assess the interventions effect on growth (LAZ, WAZ, and WLZ)

CONTACTS AND LOCATIONS:
Overall Officials: Given Chipili, Principal Investigator — Mukuba University, Kitwe, Zambia
Locations (1):
- Shikamushile Rural Health Centre, Samfya, Luapula Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
This study is part of my PhD. The information will be shared on the Stellenbosch University website two years after graduation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: Through the Stellenbosch University official website